CLINICAL TRIAL: NCT00703378
Title: Target Dosing of Docetaxel Through Pharmacokinetic/Pharmacodynamic Optimisation of the First Chemotherapeutic Cycle
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Haematology-Oncology, Dr. Goh Boon Cher, National University Hospital, Singapore
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PK01/06/05; 2005/00082 (Other: NHG Domain Specific Review Boards)
Record Dates: First submitted 2008-06-20; First posted 2008-06-23 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Solid Tumors
MeSH Terms: interventions — Docetaxel

ARMS (3):
- Group 1 (Experimental): Group 1: normal liver function
  Interventions: Drug: Docetaxel (Taxotere®)
- Group 2 (Experimental): Group 2: AST and/or ALT up to 1-5 x upper limit of normal; SAP 1- 5x upper limit of normal, total bilirubin within normal limits
  Interventions: Drug: Docetaxel (Taxotere®)
- Group 3 (Experimental): Group 3: Any SAP and AST/ALT >5-10 x upper limit of normal and/or total bilirubin 1-1.5 x upper limit of normal
  Interventions: Drug: Docetaxel (Taxotere®)

INTERVENTIONS:
Drug: Docetaxel (Taxotere®) — Phase 1 Cycle 1 and 2 Patients in group 1 receive 40mg/m2/week of docetaxel in a 1-hour infusion. Patients in group 2 receive 30mg/m2/week of docetaxel in a 1-hour infusion. Patients in group 3 receive 20mg/m2/week of docetaxel in a 1-hour infusion.
  Other Names: Taxotere®

SUMMARY:
Primary Objective

1. To develop a pharmacokinetic-pharmacodynamic (PD) model for optimisation of docetaxel dosing

Secondary Objectives

1. To establish an exposure-toxicity (neutropenia) relationship for docetaxel
2. To determine the exposure breakpoint for docetaxel toxicity based on a neutropenia PD model
3. To identify demographic, pathophysiological and/or phenotypic covariates predicting docetaxel clearance
4. To prospectively validate this PK-PD model for optimisation of docetaxel dosage and determination PK variability and toxicity

DETAILED DESCRIPTION:
Rationale

Poor tolerance of standard docetaxel dosage regimens used as a single agent in Asians has been clearly demonstrated by our group in 2 separate studies. Neutropenia emerged as the most prominent manifestation of chemotherapy toxicity [12, 20]. While this has been attributed to the lower docetaxel CL derived in our Asian patients, an optimal dosage regimen taking into account the extensive genetic polymorphisms associated with CYP3A4 has yet to be established. The use of ketoconazole as a potent CYP3A4 modulator to reduce pharmacokinetic variability of docetaxel did show >2-fold reduction in docetaxel dosage, but inter-individual variability in CL was not significantly reduced. There was also poor correlation of docetaxel CL to midazolam phenotyping of CYP3A4 with the addition of ketoconazole to the regimen [23]. Since the use of an additional modulator failed to achieve the desired reduction in pharmacokinetic variability, the idea of using low-dose docetaxel to predict its own pharmacokinetic parameters appeared feasible, safe and an appealing approach.

The more acute toxicities of docetaxel, such as neutropenia, stomatitis, neurological toxicities and fluid retention are more frequently associated with the 3 weekly than weekly dosing schedule. This study is designed so that the less toxic weekly schedule is used for PK/PD correlation. This information would be utilized to derive an optimal dosage for the 3 weekly regimen that follows since cumulative myelosuppression was not observed with previous weekly docetaxel for metastatic breast cancer [31].

Currently patients with impaired liver function manifested by elevated baseline ALT/AST more than 1.5 more than the institutional limits of normal are not treated with the recommended dose of docetaxel because of impaired clearance of docetaxel. Theoretically, these patients may benefit from docetaxel treatment, but the dose will need to be individualized based on hepatic drug clearance to avoid toxicity. To determine the clinical usefulness of our strategy of predicting docetaxel clearance and individualised dosing based on clearance and a PD model, patients with a certain extent of liver dysfunction will be included into the study. They will be divided into 3 groups according to the level of AST/ALT and SAP, total bilirubin, and initial weekly doses as well as q3weekly doses will be lower than the recommended doses for patients with normal liver function. Previous investigators have reported the feasibility of using the erythromycin breath test as an in vivo probe for CYP3A activity and docetaxel clearance in patients with liver dysfunction (Baker SD et al Evaluation of CYP3A activity as a predictor covariate for docetaxel clearance Proceedings of ASCO 2004; 128: 2006abs).

2.4 Hypothesis

The hypothesis for this study is that PK/PD guided dosing of docetaxel will reduce the variability in docetaxel PK while achieving the maximum exposure desired within acceptable limits of toxicity. At this juncture, this is a novel approach in oncology to fully exploit the potential of using low-dose docetaxel as its own probe drug to individualise and optimise dosage for subsequent chemotherapy treatment without having to use other agents to modulate or predict drug metabolism and clearance.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed malignancy that is metastatic or unresectable and for which docetaxel is indicated.
2. Patients must have measurable or evaluable disease.
3. With the exception of alopecia, fatigue, nausea and asthenia, patients must have resolution of all acute toxic effects of any prior surgery' radiotherapy or chemotherapy to National Cancer Institute (NCI) Common Toxicity Criteria version 3.0 (see Appendix A) grade < 1.
4. Patients must have ECOG performance status < 2 (Karnofsky >60%, see Appendix B).
5. Patients must have a life expectancy of greater than 3 months.
6. Patients must have normal renal and marrow function as defined below:

   * leukocytes ≥3,000/μl
   * absolute neutrophil count ≥1,500/μl
   * platelets ≥100,000/μl
   * haemoglobin ≥7g/dL
   * creatinine ≤1.5 X institutional upper limit of normal
7. Patients with abnormal liver function tests (AST/ALT ≤ 10 x institutional upper limits of normal; SAP < 5x ULN; total bilirubin ≤ 1.5x ULN) will be eligible for enrolment.
8. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Females with childbearing potential must have a negative serum pregnancy test within 7days prior to study enrollment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
9. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
2. Patients may not be receiving any other investigational agents.
3. Patients who have rapidly progressive intracranial or spinal metastatic disease (including patients who require corticosteroid for CNS disease).
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to docetaxel or other agents used in study.
5. Patients who have prior medications known to be metabolized by or induce/inhibit CYP3A4 within 1 week (see appendix C).
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Pregnant women are excluded from this study because docetaxel is embryotoxic/fetotoxic with the potential for abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with docetaxel, breastfeeding should be discontinued if the mother is treated with docetaxel. These potential risks may also apply to other agents used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2006-05; Primary Completion 2011-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
change in neutrophil counts and docetaxel AUC | 3 weeks
  . Based on maximal acceptable toxicity, expressed as the reduction in neutrophil count, the corresponding breakpoint for AUC will be identified as the PK target. Both linear regression and nonlinear mixed effects modeling will be employed to establish a relationship between docetaxel CL and demographic, phenotypic and pathophysiological factors.

SECONDARY OUTCOMES:
Pharmacokinetic sampling of docetaxel serum concentrations | 7 weeks
  Pharmacokinetic sampling of docetaxel serum concentrations will be carried out around the first course of docetaxel administration of both cycles 1a and 1b of the chemotherapy regimen. The time points elected for docetaxel sampling are: 0h (baseline), 15mins, 1.5h, 3h, 4h, 6h and 24h.

CONTACTS AND LOCATIONS:
Overall Officials: Boon Cher Goh, MBBS, MRCP, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Goh BC, Lehnert M, Lim HL, Ng AW, Chan CC, Kong HL, Lee SC, Wee J, Chua ET, Wong JE. Phase II trial of docetaxel in Asian patients with inoperable stage III non-small cell lung cancer. Acta Oncol. 2000;39(2):225-9. doi: 10.1080/028418600430824. PMID 10859016
- [Background] Goh BC, Lee SC, Wang LZ, Fan L, Guo JY, Lamba J, Schuetz E, Lim R, Lim HL, Ong AB, Lee HS. Explaining interindividual variability of docetaxel pharmacokinetics and pharmacodynamics in Asians through phenotyping and genotyping strategies. J Clin Oncol. 2002 Sep 1;20(17):3683-90. doi: 10.1200/JCO.2002.01.025. PMID 12202670
- [Derived] Syn NL, Wang L, Wong AL, Soe MY, Chuah B, Chan D, Tan SH, Soo RA, Lee SC, Goh BC, Yong WP. Dose modifications in Asian cancer patients with hepatic dysfunction receiving weekly docetaxel: A prospective pharmacokinetic and safety study. Cancer Sci. 2016 Feb;107(2):173-80. doi: 10.1111/cas.12856. Epub 2016 Feb 8. PMID 26663719